CLINICAL TRIAL: NCT04886102
Title: Molecular Epidemiology of Hepatitis B in Cayenne General Hospital, French Guiana
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier de Cayenne (Other)
Collaborators: Hospital Avicenne (Other); University Hospital, Montpellier (Other); Direction Générale de l'Offre de Soins (Other Government)
Responsible Party: Sponsor
Other Study IDs: EMOHCAY
Record Dates: First submitted 2021-01-27; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Hepatitis B, Chronic; Adults
Keywords: Hepatitis B, Chronic; Hepatitis B Virus Infection; Adults; French Guiana; Hepatitis C Virus Infection; Co-infection; Chain of transmission; Epidemiology, molecular; Viral phylodynamics; Viral phylogenetics
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B; Hepatitis C; Coinfection | interventions — Fumigant 93

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — An additional 5 mL venous blood tube taken from patients during their routine medical check-up at the hospital on which the serology and molecular biology analyzes of hepatitis B and D and the phylogenetic and phylodynamic analyzes of hepatitis B will be performed
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: An additional 5 mL venous blood tube taken from patients during their routine medical check-up at the hospital — Research protocol involving the human person (Category 3 - Non-interventional research_ not related to a health product) Serology, molecular biology, phylogenetic and phylodynamic analyzes of hepatitis B and D
  Other Names: Molecular biology analyzes of hepatitis B and D; Phylogenetic and phylodynamic analyzes of hepatitis B; Phylogenetic and phylodynamic analyzes of hepatitis C

SUMMARY:
In South America, the prevalence of HBV is variable but high (> 8%) in the Amazon basin. In some areas, a third of HBsAg carriers are also infected with HDV, a major comorbidity factor. The pre-core mutations are associated with the negative HBe Ag phenotype which is associated with a more severe course. These mutations are of increasing and high frequency. French Guiana is populated by populations of African, European and Asian origins with chains of viral transmission which are not known and viruses probably of different origins with variable virulence and transmission potentials.

DETAILED DESCRIPTION:
Human demography and migrations play a crucial role in the phylogeography of viral populations. Hepatitis B viruses are characterized by a high genetic diversity which results from the fact that this virus uses a reverse transcriptase during its replicative cycle, which induces errors and therefore variation. A dozen genotypes have so far been described and are subdivided into sub-genotypes which have a distinct ethnogeographic distribution. Genotypes A and D are ubiquitous and represent the most common genotypes in Europe; genotypes B and C are very common in Asia and Oceania, genotype E in Central Africa and West Africa, genotypes H and F in Latin America and Alaska, and Genotype I in Southeast Asia. The populations originating from these different continents are all represented in Guyana and it is therefore interesting to understand what are the chains of transmission and the phylodynamic aspects of the epidemic in French Guiana. In addition, the different genotypes have variable clinical consequences, and this in different ways depending on the ethnicity of the host. Thus, in Mexico, the F and H genotypes appear to be rather benign in the Amerindians among whom they have circulated for a long time. On the other hand, genotypes F, A and D are of rather severe evolution in Mexicans of Caucasian origin, thus suggesting that the immunogenetic factors of the host are important determinants of the pathogenic power of the viruses (Roman and al WJG 2014).

Some pre-core mutations leave the virus with the capacity to replicate. The absence of the HBe antigen deprives the immune system of an important target and the virus can therefore continue to replicate. These pre-core mutations are associated with the HBe Ag negative phenotype (7 to 30% of patients) which is associated with a more severe course of chronic hepatitis. These mutations are of increasing and high frequency (Funk ML, and al 2001).

Addiction to crack cocaine is widespread in French Guiana and appears to be one of the drivers of the epidemic. The pipes used to smoke crack cause burns on the lips and when sharing the pipe could contribute to increasing the risk of transmission (Fischer and al 2008). Risky sexual behavior is associated with the use of crack cocaine, suggesting that there may be specific chains of transmission around crack users.

Primary objective Identify the factors associated with different genotypes (age, sex, country of birth, sexual orientation, sexual risk taking, notion of IV drug addiction, crack ...) in order to identify specific chains of transmission in French Guiana.

Secondary objectives

* Describe the molecular epidemiology of hepatitis B (AgS and pre-core mutations) in French Guiana
* Carry out the phylodynamic study of the different HBV genotypes in order to reconstruct the history of the epidemic in French Guiana
* Identify the clinical prognostic factors associated with the different genotypes and phylogenetic aspects in order to identify the viruses with the greatest pathogenic potential in French Guiana
* Describe the molecular epidemiology of hepatitis D in B-D coinfected in French Guiana

Cross-sectional, monocentric, observational study with biological collection.

Research protocol involving the human person (Category 3 - Non-interventional research_ not related to a health product)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Person with confirmed chronic hepatitis B
* Person who does not object to their participation in the protocol
* HBV viral load> = 500 copies / mL
* Person who has planned / is willing to have their next HBV assessment of current care taken at the Cayenne Hospital center

Exclusion Criteria:

* Refusal to participate
* Age <18 years old
* Person opposing their participation in the protocol
* HBV viral load <500 copies / mL
* Person who has not planned / been unwilling to have their next HBV assessment of current care taken at the Cayenne Hospital center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients infected with hepatitis B followed at the Cayenne hospital center (adult day hospital consultations, consultations with the infectious and tropical diseases department and hepatology B medicine consultations)
  Estimated size of target population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-02-11 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Hepatitis B virus (HBV) sequencing | 2 years
  The mutations studied will be those relating to AgS and to the pre-core regions.
  The viral nucleic acids will be extracted using the Qiagen® technique on the Qiacube® machine. The HBV genotyping will be carried out by sequencing the nucleotides of a DNA segment amplified from the HBV S gene (nt 414 to nt 822, reference sequence HBV strain NC003977). In order to study the genetic proximity between the HBV strains, the samples will be subjected to whole genome sequencing based on the method of Ramachandran et al using two amplification steps. The first round of whole genome amplification will be followed by a second round of PCR nested on 6 overlapping fragments of 600bp each.
  A phylodynamic approach will estimate the aspects time of viral evolution. Phylogenetic trees will be produced to illustrate the genetic differences between the different types of viruses circulating in French Guiana with Mega software.

SECONDARY OUTCOMES:
Hepatitis D virus (VHD) sequencing | 2 years
  In patients also with HDV infection, HDV genotyping will be performed by nucleotide sequencing and phylogenetic analysis of the amplified R0 regions of the genome (nt 889 to nt 1289). The complete sequences will be characterized by the amplification and sequencing of 4 overlapping regions covering the entire genome: R0 (nt 889 to nt 1289), R1 (nt 320 to nt 1289), R2 (nt 889 to nt 420) and R3 (nt 200 to nt 560).
  A phylodynamic approach will estimate the aspects time of viral evolution. Phylogenetic trees will be produced to illustrate the genetic differences between the different types of viruses circulating in French Guiana with Mega software.
Liver function Markers | 2 years
  Various liver function markers will be taken. Several groups will be distinguished and compared in terms of genotype and subclades, thus testing the null hypothesis of an absence of difference between genotypes and markers of evolution. Association will be assessed using Chi square tests for crosstabulation of categorical variables and other genotypes (exploratory analyses).

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu NACHER, MD, PhD, Principal Investigator — Centre Hospitalier de Cayenne
Locations (1):
- General Hospital of Cayenne, Cayenne, French Guiana